CLINICAL TRIAL: NCT04421287
Title: Clinical Study on the Effect of Zhenyuan Capsule on Cardiopulmonary Function in Patients With Stable Coronary Heart Disease With Qi Deficiency and Blood Stasis
Brief Title: Clinical Study on the Effect of Zhenyuan Capsule on Cardiopulmonary Function in Patients With SCAD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xiyuan Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020XLA018-2
Record Dates: First submitted 2020-05-06; First posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-04

CONDITIONS: Stable Coronary Heart Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double mind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zhenyuan capsule (Experimental)
  Interventions: Drug: Zhenyuan capsule
- Zhenyuan capsule placebo (Placebo Comparator)
  Interventions: Drug: Zhenyuan capsule

INTERVENTIONS:
Drug: Zhenyuan capsule — 0.25g/ tablets, 2 tablets / TID, for 12 weeks

SUMMARY:
A randomized, double-blind, placebo trial was adopted, and cardiopulmonary exercise load test (CPET) was used to detect peak oxygen uptake (PeakVO2) and exercise metabolic equivalent (METs) to confirm the clinical effect of Zhenyuan capsule on improving cardiopulmonary endurance in patients with coronary heart disease of qi deficiency and blood stasis.

ELIGIBILITY:
Inclusion Criteria:

* Results of coronary angiography or spiral CT:Patients with coronary artery stenosis ≥ 50%, or with a clear history of myocardial infarction, or stable condition more than one month after ACS treatment (percutaneous coronary intervention therapy, PCI, coronary artery bypass graft, CABG)；
* LVEF≥40%；
* Angina grade Ⅰ-Ⅱ (CCS grade);
* The syndrome differentiation of traditional Chinese medicine is the syndrome of qi deficiency and blood stasis；
* 18 years old ≤ age ≤ 75 years old；
* In accordance with the risk stratification of cardiac rehabilitation in patients with coronary heart disease, the patients with moderate and low risk can carry out cardiopulmonary rehabilitation by exercise；
* Those who sign the informed consent form.

Exclusion Criteria:

* Patients with acute myocardial infarction or unstable angina pectoris, or within one month after PCI or CABG;
* Patients with absolute and relative contraindications in accordance with cardiopulmonary exercise test;
* Patients who took Zhenyuan capsule in the past 1 month or participated in other clinical trials in the past 1 month；
* Renal insufficiency, serum creatinine > 2.5mg / dl in male and > 2.0mg/dl in female；
* Patients with obvious liver disease or both ALT and AST were 3 times higher than the normal upper limit；
* New York heart function (NYHA) grade IV, or patients with recurrent malignant arrhythmias;
* Complicated with chronic obstructive pulmonary disease or even respiratory failure, or complicated with pulmonary infection;
* Diabetic patients with random blood glucose ≥ 13.7mmol/L or glycosylated hemoglobin ≥ 9.5%;
* Pregnant or preparing pregnant women, lactating women;
* Patients with acute cerebrovascular diseases; malignant tumors or patients with life expectancy of less than 1 year; patients with severe hematopoietic diseases; patients with severe mental illness;
* For those who are allergic to the known ingredients of the drug.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Cardiopulmonary function index change | Change from Baseline VO2 peak at 12 weeks / 16 weeks after drug treatment;
  Peak Oxygen Uptake（Peak VO2）；Heart rate、Stroke volume and arteriovenous oxygen difference will be combined to report VO2 peak in mL/kg/min(milliliters of oxygen per kilogram of body weight per minute )；

CONTACTS AND LOCATIONS:
Overall Officials: Long C Wang, doctorate, Study Chair — Xiyaun Hospital of China Academy of Chinese Medical Sciences
Locations (1):
- Xiyuan Hospital of China Academy of Chinese Medical Sciences, Beijing, China